CLINICAL TRIAL: NCT06898697
Title: Midazolam or Fentanyl as Adjuvants to Epidural Bupivacaine Plus Dexamethasone for Analgesia After Lumbar Spine Fixation: A Randomized Clinical Study
Brief Title: Midazolam or Fentanyl as Adjuvants to Epidural Bupivacaine Plus Dexamethasone for Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Marwa Mohamed Medhat, assistant professor of anesthesia and surgical intensive care (Principal Investigator), Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZU-IRB#1075/ 25-Feb-2025
Record Dates: First submitted 2025-03-13; First posted 2025-03-27 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Lumbar Spine Fixation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fentanyl (Active Comparator): Patients will receive 10 ml of bupivacaine 0. 25 % plus 100µg fentanyl in 2ml plus 2ml (8mg) dexamethasone (14 ml total volume).
  Interventions: Drug: Epidural fentanyl
- midazolam (Active Comparator): Patients will receive 10 ml of bupivacaine 0.25 % plus 2mg midazolam in 2ml plus 2 ml (8mg) dexamethasone with (14 ml total volume).
  Interventions: Drug: epidural midazolam

INTERVENTIONS:
Drug: Epidural fentanyl — Fentanyl will be injected in the epidural space by the surgeon one or two levels above the surgical site.
  Arms: fentanyl
Drug: epidural midazolam — midazolam will be injected in the epidural space by the surgeon one or two levels above the surgical site.
  Arms: midazolam

SUMMARY:
The purpose of this study is to compare better postoperative analgesia after lumbar spine Fixation using either epidural bupivacaine with midazolam or fentanyl with the combination of dexamethasone.

DETAILED DESCRIPTION:
After being informed about the study and potential risks. A computer-generated randomization table will randomize all patients giving written consent into 2 groups, each containing 51 patients. In the Fentanyl Group :.Patients will receive 10 ml of bupivacaine 0. 25 % plus 100µg fentanyl in 2ml plus 2ml (8mg) dexamethasone.In Midazolam Group: Patients will receive 10 ml of bupivacaine 0.25 % plus 2mg midazolam in 2ml plus 2 ml (8mg) dexamethasone

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from the patient.
* Physical status: ASA 1& II.
* BMI = (25-30 kg/m2).
* Type of operation: elective lumbar spine Fixation.

Exclusion Criteria:

* Altered mental state.
* Patients with known history of allergy to study drugs.
* Advanced hepatic, renal, cardiovascular, and respiratory diseases.
* Patients with chronic pain.
* Contraindications of regional anesthesia, e.g., allergy to local anesthetics, coagulopathy, or septic focus at site of injection.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
the time to first call to rescue analgesia (ketorolac) | day 1

SECONDARY OUTCOMES:
The Numerical Pain Rating Scale | 24 hours postoperative]
  A ten-centimeter Numerical Pain Rating Scale (0 - no pain and 10 - worst pain)
The total postoperative opioid consumption in the first 24 hours. opioid consumption | 24 hours postoperative
the duration of hospital stay | up to 1 week
  from the post operative day till discharge from hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine,Zagazig University, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No